CLINICAL TRIAL: NCT05687019
Title: Efficacy of Hyaluronic Acid and Chondroitin Sulphate in Intravesical Injections on Functional Recovery After Holmium Laser Surgery for Prostate Adenoma (HOLEP-AHCS)
Brief Title: Efficacy of Hyaluronic Acid Injections on Functional Recovery After Surgery for Prostate Adenoma
Acronym: HOLEP-AHCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-A01882-41
Record Dates: First submitted 2023-01-06; First posted 2023-01-17 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Prostatic Adenoma
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient undergoing prostate enucleation by Holmium Laser (Experimental): It is based on a pulsed laser at a wavelength of 2140 nm, which penetrates the tissues over a very short distance. The prostate tissue must therefore be in contact with the laser fiber to be cut or vaporized, and hemostasis will take place nearby. The procedure lasts approximately one hour.
  Interventions: Combination Product: Intravesical instillations of Ialuril® Prefill

INTERVENTIONS:
Combination Product: Intravesical instillations of Ialuril® Prefill — 5 injections of Ialuril® Prefill on D0 or D1, D7, D14, D21 and D28 after Holmium laser surgery for prostate adenoma

SUMMARY:
The purpose of this study is to evaluate the score on urinary function (International Prostate Score Symptom) at 28 days.

The main objective is to assess the efficacy of treatment with Ialuril® Prefill on functional recovery at 4 weeks, based on the International Prostate Score Symptom.

A paired test will be performed to compare the International Prostate Score Symptom score between 0 and 28 days.

DETAILED DESCRIPTION:
This is an interventional, non-comparative, open-label, monocentric study aimed at evaluating treatment with hyaluronic acid in patients who have undergone surgery (HOLEP procedure) for prostatic adenoma.

ELIGIBILITY:
Inclusion Criteria:

* Patient eligible for a HOLEP procedure, according to the investigator ;
* Patient able to understand the information related to the clinical investigation, to read the information leaflet and agrees to sign the consent form.

Exclusion Criteria:

* Known intolerance to one of the treatment components: hyaluronic acid, chondroitin sulphate, calcium chloride;
* Prostatic volume greater than 140 cm3;
* Patient under anticoagulant treatment for secondary prevention;
* Patient under guardianship or curatorship, or under a regime of deprivation of liberty;
* Participating patient, or in a period of exclusion from another clinical trial;
* Patient not benefiting from a social security scheme.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-09-12 (Actual); Primary Completion 2025-06-24 (Actual); Study Completion 2025-06-24 (Actual)

PRIMARY OUTCOMES:
International Prostate Score Symptom on Day 28 | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique La Croix du Sud, Quint-Fonsegrives, France

IPD SHARING:
Plan to Share IPD: No